CLINICAL TRIAL: NCT06698692
Title: Real-world Assessment of Trilaciclib for the Prevention of Chemoradiotherapy-Induced Myelosuppression in Esophageal Squamous Cell Carcinoma
Brief Title: Trilaciclib for the Prevention of Chemoradiotherapy-Induced Myelosuppression in Esophageal Squamous Cell Carcinoma
Acronym: COSELA
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: COSELA-ESCC-02
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: ESCC
Keywords: trilaciclib
MeSH Terms: interventions — trilaciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Unsaved Biospecimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group: Trilaciclib combined with chemoradiotherapy
  Interventions: Drug: Trilaciclib Injection [Cosela]
- Control group: chemoradiotherapy

INTERVENTIONS:
Drug: Trilaciclib Injection [Cosela] — Trilaciclib Combined chemoradiotherapy
  Groups: Observation group

SUMMARY:
Clinical data of patients with synchronous radiotherapy for esophageal cancer in the Department of Radiology of Jiangsu Provincial People's Hospital were collected. Patients were divided into trilaciclib group (34 cases) and control group (169 cases) based on whether trilaciclib was used or not. Patients in the trilaciclib group were given trilaciclib before each chemotherapy treatment. Propensity score matching (PSM) was used to balance the baseline characteristics between the two groups on a 1:1 ratio. After pairing, the rates of bone marrow suppression and other adverse events were compared between the two groups.

DETAILED DESCRIPTION:
chemoradiotherapy-induced myelosuppression (CIM) is the most common adverse event of concurrent chemoradiotherapy for esophageal cancer, often leading to reduction, delay or even cessation of chemotherapeutic agents. Clinical treatments for CIM mainly include various hematopoietic growth factors and blood transfusion. However, these interventions target only a single spectrum of blood cells and are susceptible to concomitant adverse events such as bone pain, thrombosis, and fever. Trilaciclib is a potent, transient, reversible CDK4/6 inhibitor and is the world's first innovative drug with lineage-wide myeloprotective effects. Its use in esophageal cancer has not been reported yet. In this study, we investigated the clinical efficacy and safety of trilaciclib in preventing myelosuppression in concurrent chemoradiotherapy for esophageal cancer for the first time.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* pathological diagnosis of esophageal squamous cell carcinoma;
* failure to undergo surgical treatment;
* completion of definitive chemoradiotherapy or chemoradiotherapy combined with immunotherapy.

Exclusion Criteria:

* history of other malignant tumors;
* difficulty in follow-up;
* insufficient clinical information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal squamous carcinoma who received concurrent chemoradiotherapy with or without trilaciclib.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥3 neutropenia | during Trilaciclib plus chemotherapy assessed up to 1 years
  Incidence of grade ≥3 neutropenia

SECONDARY OUTCOMES:
Incidence of Adverse Events | during Trilaciclib plus chemotherapy assessed up to 1 years
  The incidence of Adverse Events according to Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Xiao L Ge, PHD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No